CLINICAL TRIAL: NCT03993834
Title: Palmar Arch Insufficiency as a Risk Factor for Radial Artery Occlusion After Transradial Catheterization - a Single-Centre Observational Study
Brief Title: Palmar Arch Insufficiency as a Risk Factor for Radial Artery Occlusion After Transradial Catheterization
Acronym: PAIRAO
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00622
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease
Keywords: Transradial catheterization; Transradial access; Radial artery occlusion; Palmar arch collateral circulation; Collateral flow index
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal modified Allen Test: Patients undergoing transradial coronary angiography with a modified Allen-Test ≤ 15 seconds
- Abnormal modified Allen Test: Patients undergoing transradial coronary angiography with a modified Allen-Test > 15 seconds

SUMMARY:
Transradial access (TRA) is commonly used in different medical fields due to the superficial position of the radial artery and related advantages. Despite its popularity, the incidence and importance of related complications, in particular, radial artery occlusion (RAO) remains unclear. Further, the only known independent predictors of the radial artery occlusion are the periprocedural anticoagulation as well as the catheter size. The effect of a variable arterial anatomy has so far not been evaluated.

In this context, most institutions prefer to evaluate the collateral circulation of the hand, i.e., the arterial palmar arch and forearm circulation before TRA. The most commonly employed tests are the modified Allen test (MAT) or the combination of pulse oximetry and plethysmography according to Barbeau.In addition, there are more precise, but still semi-quantitative non-invasive methods for palmar arterial collateral function testing.

Despite the wealth of these variably accurate and practical tests, invasive and direct hemodynamic measurement of the arterial forearm circulation and its components is lacking. Thus, the human physiologic circulatory reference at this site has been unknown so far. Further, the need of pre-procedural testing itself can be questioned in light of the reported, widely varying prevalence of RAO (1-38%) or critical ischemia (0-0.09%) after TRA.

The present study investigated in a first step the invasively obtained, pressure-derived hemodynamic function, i.e., the physiology of the human arterial palmar arch and forearm collateral circulation and in a second step the clinical consequences of the variable palmar arterial anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient receiving transradial coronary angiography and undergoing evaluation of the palmar arterial arch circulation as a quality control
* Written informed consent to participate in the follow-up Doppler ultrasound examination

Exclusion Criteria:

* Changed anatomical conditions of the radial artery, e.g. after coronary artery bypass surgery with radial harvest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients electively referred for coronary angiography undergoing transradial access
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | 3 months after transradial coronary angiography
  Frequency of radial artery occlusion after transradial coronary angiography; assessed by Doppler ultrasound measurements

SECONDARY OUTCOMES:
Palmar arch collateral circulation | Measured during transradial access of the coronary angiography, expected to be 1 minute after local anesthesia and direct after successful punctuation of the radial artery
  Quantitatively measure of the pressure-derived function of the palmar collateral circulation during transradial catheterization. Assessment of the collateral function by setting the invasively obtained blood pressure during external occlusion in relation to the unaffected blood pressure of the radial artery.
Radial artery stenosis | 3 months after transradial coronary angiography
  Frequency of radial artery stenosis after transradial coronary angiography; assessed by Doppler ultrasound measurements

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- University Hospital Inselspital, Bern, Bern, Switzerland

REFERENCES:
- [Derived] Bigler MR, Buffle E, Rappo MV, Grossenbacher R, Tschannen C, Seiler C. Association of Palmar Arch Collateral Function and Radial Artery Occlusion After Transradial Access. Am J Cardiol. 2022 Apr 1;168:151-158. doi: 10.1016/j.amjcard.2021.12.020. Epub 2022 Jan 20. PMID 35065801
- See also: Jolly SS et al. Lancet 2011 - Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. — https://www.ncbi.nlm.nih.gov/pubmed/21470671